CLINICAL TRIAL: NCT04947865
Title: Characterization of Abnormal Reflex Couplings Via H-reflex Stimulation
Brief Title: Reflex Excitability in Post-stroke Stiff-Knee Gait
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Sulzer, Associate Professor, Department of Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-01-0022; R01HD100416 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-07-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Chronic Stroke; Gait, Hemiplegic; Gait, Spastic; Gait Disorder, Sensorimotor; Gait Disorders, Neurologic; Walking, Difficulty
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Post-stroke Stiff-Knee Gait Participants (Experimental): Individuals with post-stroke Stiff-Knee gait
  Interventions: Other: Peripheral nerve stimulation
- Healthy Individuals (Experimental): Healthy Individuals
  Interventions: Other: Peripheral nerve stimulation; Device: Commercial knee brace

INTERVENTIONS:
Other: Peripheral nerve stimulation — Electrical stimulation of peripheral nerves to measure resulting gait kinematics and surface muscle activity
Device: Commercial knee brace — Knee brace used to limit knee mobility in healthy individuals to imitate stroke survivors and measure resulting gait kinematics and surface muscle activity.
  Arms: Healthy Individuals

SUMMARY:
The purpose of this study is to examine the reflex excitability of the rectus femoris in individuals with and without post-stroke Stiff-Knee gait. We use electrical stimulation of the peripheral nerve innervating the rectus femoris for a well-controlled reflex stimulus. We are investigating whether reflex excitability of the rectus femoris correlates with gait kinematics.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the role of hyperreflexia in post-stroke Stiff-Knee gait function. In one aim,

ELIGIBILITY:
Inclusion criteria:

* Aged at least 18
* Premorbidly independent
* If post-stroke, mild to moderate impairment determined by standard practices per the physical therapist
* Able to continuously walk for 30 minutes
* If post-stroke, reduced knee flexion during walking relative to unimpaired side
* If post-stroke, hemiparesis
* Ability to provide informed consent

Exclusion criteria:

* No history of serious lower limb musculoskeletal injury
* No functionally relevant osteoarthritis and weight-bearing restrictions
* No functionally relevant polyneuropathy
* No functionally relevant cognitive impairment
* No functionally relevant vision impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Surface electromyographic recording of leg muscles during different conditions | 1 hour
  Recording electrical activity of leg muscles during walking in response to peripheral nerve stimulation

SECONDARY OUTCOMES:
Circumduction measure | 1 hour
  Hip abduction joint motion measured with motion capture

CONTACTS AND LOCATIONS:
Overall Officials: James S Sulzer, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States